CLINICAL TRIAL: NCT02677675
Title: Effectiveness of Mobile Phone Technology in Improving Adherence and Treatment Outcomes Among HIV Positive Patients on Antiretroviral Therapy (ART) in Malaysia
Brief Title: Effectiveness of Mobile Phone Technology on Adherence and Treatment Outcomes Among HIV Positive Patients on ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr. Surajudeen Abiola Abdulrahman, Graduate Researcher, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UPM/TNCPI/RMC/1.4.18.1 (JKEUPM
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: HIV
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (reminder module) (Experimental): A "reminder module" which included standardized weekly SMS medication reminders (sent at 9am every Monday); SMS reminder 3 days prior to scheduled clinic appointments (individualized and sent at lunch time), and an average of 90sec lunch hour telephone call reminders a day prior to scheduled clinic appointment (in addition to standard care - routine adherence counselling) was delivered consistently for 24 weeks to respondents in the intervention group by two trained PLHIV (research assistants)
  Interventions: Behavioral: Intervention (reminder module)
- Control (standard care) (No Intervention): Control group received standard care only (routine adherence counselling and paper-based appointment scheduling)

INTERVENTIONS:
Behavioral: Intervention (reminder module) — Reminder module (delivered via SMS and telephone call reminders)
  Arms: Intervention (reminder module)

SUMMARY:
The objective of this study was to determine the effectiveness of mobile phone technology (SMS and telephone call reminders) in improving adherence and treatment outcomes among HIV positive patients on ART in Malaysia.

DETAILED DESCRIPTION:
This study was a 2 arm, parallel group, randomized single blind clinical trial involving 242 randomly selected and allocated adult Malaysian HIV positive patients who were enrolled into Antiretroviral Therapy (ART) care at Infectious Disease Clinic of Hospital Sungai Buloh, Malaysia. Recruitment commenced in January 2014 and follow up ended in December 2014. Each individual patient was followed up for a period of 6 months on ART. A reminder module (delivered via Short Message Service (SMS) and telephone call reminders) was developed based on the Theory of Planned Behavior. The reminder module which included standardized weekly SMS medication reminders (sent at 9am every Monday); SMS reminder 3 days prior to scheduled clinic appointments (individualized and sent at lunch time), and an average of 90sec lunch hour telephone call reminders a day prior to scheduled clinic appointment (in addition to standard care - routine adherence counselling) was delivered consistently for 24 weeks to respondents in the intervention group by two trained PLHIV (research assistants) while respondents in the control group received standard care only. Each patient in the intervention group had a minimum of three (during clinic visits at month 1, month 3 and month 6) individual counselling sessions with the research assistants lasting an average of 15 minutes per encounter. To ensure confidentiality, typical medication reminder text messages included a short slogan in Malay language "Apa khabar" "Ini untuk menberithau anda ubat" meaning "How are you?" "This is to remind you of your medications". Appointment reminder text message was "Apa khabar" "Tolong ingat tarikh temu janji lusa" meaning "How are you?" "Remember your appointment day after tomorrow" and telephone conversation was standardized and short, with the message "Apa khabar" "Tolong ingat tarikh temu janji besok" meaning "How are you?" "Remember your appointment tomorrow". Patients were not required to provide any responses to the text messages. However, a log of text message communications and telephone calls was recorded and kept.

Upon enrollment and randomization to a treatment arm, baseline data on socio-demographic factors, clinical symptoms and adherence behavior of respondents was collected using modified, pre-validated, reliable, self-administered Adult AIDS Clinical Trial Group (AACTG) adherence questionnaire. The baseline medication adherence questionnaire consisting of nine sections was used to collect data on patient's understanding and level of preparedness to take HIV medications, level of psychosocial support from their friends and families, reasons for missing medications as well as period and number of missed medications. Other information collected were on patient's psychosocial symptoms and well-being, history of drug and alcohol use, socio-demographic characteristics, source of HIV infection and disclosure status, and review of their symptoms in the past 30 days. Responses to questions in sections A - E1 were graded on a 4-point Likert scale, sections E2 and I on a 5-point Likert scale, section F on a multiple scale (multiple choice, 2-point and 4-point scales), H on a 2-point scale, while section G had 5 questions on socioeconomic and demographic characteristics.

Baseline weight, blood pressure, CD4 count, Viral load, as well as results of renal profile and liver function tests were also collected and recorded.

Adherence measurement was repeated at 3 and 6 months follow-up using self-administered AACTG follow-up adherence questionnaires which consisted of eight sections (sections A - H) and a total of 49 questions graded on a combination of Likert and "Yes" or "No" scales, used for assessing how well the patient has adhered to their medications and specific instructions about their regimen within the past 3 months, with particular emphasis on the past four days. It also contained a review of their symptoms during the past four weeks as well as their current TB status and OI index. Section A consisted of a review of the respondent's current medications, by evaluating their understanding and knowledge of the treatment regimen in terms of drug name, frequency and strength of dosage, how long the patient has been on the regimen, number of pills per dose as well as number of doses missed in the past four days. This section was completed in a collaborative manner between the study personnel and the patient. Responses to questions in sections B, C, D & H were graded on a 5-point Likert scale, E on a 2-point scale, F on a 6-point scale, and G on a 4-point scale.

CD4 count, viral load, weight, full blood count, liver function, renal profile and blood pressure measurements were repeated at 6 months follow-up period, and the results retrieved from laboratory records.

Adherence scores were calculated using a standardized adherence index formula adopted from Reynolds et al.(2007). Data on regularity of respondents' scheduled clinic visits was obtained by the research assistants (for whom access was duly sought and provided by the hospital management) from the hospital's electronic medical records system using standardized data extraction forms and corroborated with drug refill appointments from pharmacy records. The research assistants accessed and recorded onto the data extraction forms, information on patient's TB status, opportunistic infection (OI) index and body weight from clinicians' notes in the electronic medical record system. Data extraction forms were reviewed periodically for completeness, correctness and accuracy by the site study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* All HIV positive patients aged 15 - 65 years, assessed and eligible for ART commencement.
* All ART eligible patients who have valid telephone numbers and can read text messages.

Exclusion Criteria:

* All HIV positive patients already commenced (current) or restarting ART due to previous default and/or lost-to-follow-up status
* Pregnant HIV-positive ART patients
* Foreigners

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Adherence (improved scheduled clinic attendance and medication adherence self-report) | Change from baseline adherence at 3 months and at 6 months
  Medication adherence was measured based on adherence ratio (for each of the 4 days prior was calculated as 1 minus (number of doses missed for the day/number of doses prescribed); adherence index based on formula adapted from Reynolds et al, 2007; and adherence category (>95% = Good adherence; 80-95% = Fair adherence; and <80% = Poor adherence) (WHO 2005).
  Scheduled clinic attendance was measured and categorized based on the number of scheduled clinic visits attended, number of times defaulted and whether or not the patient was lost-to-follow-up
  (a) Regular clinic attendee - a person who has never missed any scheduled clinic appointment (b) Defaulter - a person who has missed one or more scheduled clinic appointment, for any reason(s) (c) Lost-to-follow-up - a person is said to be lost to follow up if s/he refuses to show up for scheduled clinic visit for 3 consecutive months, after 3 consecutive attempts to track the client and bring them back on treatment.

SECONDARY OUTCOMES:
Immunological (improved CD4 count) | Change from baseline CD4 count at 6 months
  cells per millimeter cube of blood
Virological (decreased viral load) | Change from baseline viral load at 6 months
  absolute counts and log10 values. Viral suppression: (a) All clients with viral load <400 copies/mL at 6 months were termed to have achieved viral suppression, and (b) viral load >400 copies/mL at 6 months was termed unsuppressed viral load.
Clinical (Improved weight) | Change from baseline weight at 6months
  weight in Kg
Clinical (TB status) | Change from baseline TB status at 6 months
  TB status: (a) No signs and symptoms of TB (b) TB suspected clinically and referred for evaluation (c) Currently on INH Prophylaxis (IPT) (d) Currently on TB treatment. This was extracted onto the AACTG questionnaires from clinician's records based on clinical evaluation during hospital visits. Patient's susceptibility to, or recovery from TB was expected to correlate with immune status/recovery
Clinical (Opportunistic infection index) | Change from baseline Opportunistic Infection (OI) index at 6 months
  OI index: (a) WHO Clinical Stage 1 (b) WHO Clinical Stage 2 (c) WHO Clinical Stage 3 (d) WHO Clinical Stage 4. This was extracted onto the AACTG questionnaires from clinician's records based on clinical evaluation during hospital visits. Patient's susceptibility to, or recovery from OIs was expected to correlate with immune status/recovery

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Study Protocol — http://www.nmrr.gov.my